CLINICAL TRIAL: NCT06230263
Title: A Comparative Study on Functional Vision in Astigmatic Patients: DAILIES TOTAL1 Toric Contact Lenses vs. Spherical Equivalent Contact Lenses in Asian Eyes
Brief Title: Comparative Functional Vision Outcomes: DAILIES TOTAL1 Toric vs. Spherical Lenses in Asian Astigmatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mopsy Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: #IIT89779909
Record Dates: First submitted 2024-01-11; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Comparative Effectiveness Research
Keywords: Astigmatism; Toric Contact Lenses; Contact Lens Satisfaction; Digital Device Usage
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: This study will follow a double-masked randomized crossover design [10], where participants will be fitted with DAILIES TOTAL1® for Astigmatism and DAILIES TOTAL1® Spherical Contact Lenses in a randomized order. Each participant will use both types of lenses over different periods.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization:
  Generate a random list of 39 labels ("A" for DAILIES TOTAL1® for Astigmatism, "B" for Spherical Contact Lenses) using a computer.
  Randomize the list order and apply matching coded stickers to lens packages. A designated unmasked examiner has exclusive access to the decoding key and does not partake in direct participant interaction or data handling.
  Visit 1:
  Confirm participant eligibility, then the unmasked examiner uses the random list to provide the coded lens package to the masked examiner.
  The masked examiner fits the participant with the first set of lenses, unaware of the type.
  Visit 3:
  The unmasked examiner repeats Visit 1's procedure for the second set of lenses. Blinded study conditions are maintained as the masked examiner fits the second pair of lenses.
  End of Study:
  The unmasked examiner decodes the lens order for data analysis. This method ensures a double-blind crossover design, minimizing bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAILIES TOTAL1® for Astigmatism (Experimental): DAILIES TOTAL1® for Astigmatism
  Interventions: Diagnostic Test: Visual acuity test
- Spherical Contact Lenses (Active Comparator): DAILIES TOTAL1® Spherical Contact Lenses
  Interventions: Diagnostic Test: Visual acuity test

INTERVENTIONS:
Diagnostic Test: Visual acuity test — Assess near high-contrast visual acuity (40cm) using EyeChart PRO on an iPad.
  Use the MNREAD app to measure:
  Reading Acuity: Smallest font size read without errors. Critical Print Size: Smallest font size for peak reading speed. Maximum Reading Speed: Time to read comfortable font size, in words per minute. Reading Accessibility Index: Single metric summarizing visual access to print. Assess near visual function with the Near Activity Visual Questionnaire.
  Evaluate distance visual acuity, both high and low contrast, using logMAR and the E-ETDRS (NIDEK SC-2000).
  Other Names: Reading acuity test; Near Activity Visual Questionnaire

SUMMARY:
The goal of this comparative clinical trial is to assess the effectiveness of DAILIES TOTAL1 Toric Contact Lenses compared to Spherical Equivalent Contact Lenses in improving the functional vision of astigmatic patients, with a particular focus on Asian individuals who frequently use digital devices.

The main questions it aims to answer are:

How do DAILIES TOTAL1 Toric Contact Lenses affect the quality of vision in daily activities, especially when using digital screens, compared to Spherical Equivalent Contact Lenses?

What is the level of comfort and overall satisfaction among participants using DAILIES TOTAL1 Toric Contact Lenses versus those using Spherical Equivalent Contact Lenses?

Participants will be asked to wear both types of contact lenses for a specified period. During this time, they will perform various tasks involving digital screens. Their vision quality and comfort levels will be monitored and recorded. They will also be asked to report their satisfaction with each type of lens and any differences in their experience with screen use.

DETAILED DESCRIPTION:
Background:

In today's digital age, individuals spend a significant amount of time using digital devices [1]. This is notably challenging for individuals with astigmatism, a condition that can impair visual acuity when using these devices [2]. Despite the prevalence of astigmatism, toric contact lens technology, which can potentially improve visual acuity for these individuals, remains underused [3][4]. Many eye care practitioners opt for spherical lenses due to perceived complexities of fitting and considerations of cost-effectiveness [5][6].

DAILIES TOTAL1® for Astigmatism contact lenses, the first and only daily disposable Water Gradient toric contact lenses, can potentially address this issue. These lenses represent a significant innovation in toric contact lens technology, offering a unique combination of breathability and exceptional comfort. The lenses utilize Water Gradient Technology, creating a gradual transition in water content from the core to the surface of the lens, with the water content approaching 100% at the lens surface. This technology enables these lenses to offer a combination of high breathability and exceptional comfort.

Unmet Medical Need:

Although toric lenses, including DAILIES TOTAL1® for Astigmatism, have been shown to improve visual acuity in astigmatic patients, their impact on real-world visual performance, particularly when using digital devices, is less understood [1]. Additionally, while many practitioners gravitate towards spherical lenses, astigmatic patients could greatly benefit from the comfort and visual acuity provided by DAILIES TOTAL1® for Astigmatism contact lenses.

Gaining insights into the real-world visual performance of astigmatic patients when using DAILIES TOTAL1® for Astigmatism contact lenses could provide valuable information to eye care practitioners and patients. This could potentially encourage the broader adoption of DAILIES TOTAL1® for Astigmatism contact lenses, improving the visual experience for astigmatic patients and addressing an unmet medical need.

Scientific Rationale:

Previous clinical studies have demonstrated the benefits of toric contact lenses in improving visual acuity in astigmatic patients[5]. However, these studies primarily used traditional high-contrast, high-luminance visual acuity testing, which may not accurately reflect the visual demands of real-world tasks, especially those involving digital devices [7][8].

DAILIES TOTAL1® for Astigmatism contact lenses stand out due to their unique Water Gradient Technology and Precision Balance 8|4® Lens Design. The gradual transition in water content from the core to the surface of the lens, with the water content approaching 100% at the lens surface, enables a combination of high breathability and exceptional comfort. The lens design ensures a quick and stable fit, with 99% first-lens fit success. Additionally, these lenses feature SmarTears® Technology, which releases an ingredient found naturally in tears to stabilize the lipid layer of the tear film, further promoting comfort for the wearer.

This study seeks to extend previous findings by evaluating the impact of DAILIES TOTAL1® for Astigmatism Contact Lenses on subjective and objective visual performance outcomes in astigmatic patients using digital devices [9]. This will involve the use of advanced digital real-world and patient-reported outcome tools, providing a comprehensive evaluation of vision beyond acuity alone. The goal is to ascertain whether the unique benefits of DAILIES TOTAL1® for Astigmatism Contact Lenses translate to improved functional vision and overall satisfaction for astigmatic patients.

Objective:

This study aims to assess the impact of DAILIES TOTAL1® for Astigmatism Contact Lenses on the functional vision of astigmatic patients as compared to DAILIES TOTAL1® Spherical Contact Lenses, using digital real-world and patient-reported outcome tools in Asian Eyes.

Hypothesis:

DAILIES TOTAL1® for Astigmatism Contact Lenses will improve both subjective and objective visual performance in astigmatic patients using digital devices compared to DAILIES TOTAL1® Spherical Contact Lenses in Asian Eyes.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Asian, confirmed through both self-report and observation by the Principal Investigator (PI).
* Age between 18 and 39 years.
* Vertexed corrected sphere power ranging from -0.50 to -6.00 diopters (D).
* Vertexed refractive cylinder power ranging from -0.75 to -1.50 diopters (D).
* Best corrected visual acuity of 20/25 or better in each eye.
* Habitual soft contact lens wear for at least 6 months and must be successfully fitted with both DT1 Spherical and Toric contact lenses.

Exclusion Criteria:

* Any history of ocular pathology or surgery.
* Presence of active ocular infection or clinically significant ocular inflammation.
* Presence of any significant binocular vision abnormalities.
* Use of gas-permeable contact lenses within 3 months prior to the study.
* Pregnancy or lactation, confirmed by self-report.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Near high-contrast visual acuity (40cm) | Day 4, Day 8
  Assess near high-contrast visual acuity (40cm) using EyeChart PRO on an iPad.

SECONDARY OUTCOMES:
Reading Acuity | Day 4, Day 8
  Reading Acuity refers to the smallest font size at which text can be read without errors.
  The MNREAD app will be used to determine the Reading Acuity, which will be reported in units of point size (pt).
Critical Print Size | Day 4, Day 8
  Critical Print Size is the smallest font size at which the individual achieves their peak reading speed.
  The MNREAD app will measure the Critical Print Size and report it in point size (pt).
Maximum Reading Speed | Day 4, Day 8
  Maximum Reading Speed is the fastest rate at which text in a comfortable font size can be read.
  The MNREAD app will record the Maximum Reading Speed in words per minute (wpm).
Reading Accessibility Index | Day 4, Day 8
  Reading Accessibility Index is a single metric that summarizes an individual's visual access to print.
  The MNREAD app will calculate the Reading Accessibility Index based on a combination of the above measures. The index will be dimensionless but will take into account the variations in font size (pt) and reading speed (wpm) to provide a standardized score reflecting overall reading accessibility.
Near Activity Visual Questionnaire (NAVQ) | Day 4, Day 8
  The Near Activity Visual Questionnaire (NAVQ) is used to assess the near visual function, which includes the ability to perform activities that require close-up vision.
  Participants will respond to the NAVQ, which will be scored on a scale ranging from 0 to 3 for each item.
  * **Scale Range**: The scale ranges from 0 to 3, where:
  * '0' indicates no difficulty,
  * '1' indicates mild difficulty,
  * '2' indicates moderate difficulty,
  * '3' indicates extreme difficulty.
  The total NAVQ score is calculated by summing the individual scores for each item. The minimum score is '0', which would indicate no difficulty with near visual tasks, and the maximum possible score is dependent on the number of items in the questionnaire.
  Lower Scores Represent**: A better outcome, with less difficulty in near visual tasks.
  Higher Scores Represent**: A worse outcome, with greater difficulty in near visual tasks.
Distance visual acuity | Day 4, Day 8
  Evaluate distance visual acuity, both high and low contrast, using logMAR and the E-ETDRS (NIDEK SC-2000).

CONTACTS AND LOCATIONS:
Overall Officials: MANKI CHAN, Principal Investigator — Mopsy Research
Locations (1):
- Mopsy Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young G, Sulley A, Hunt C. Prevalence of astigmatism in relation to soft contact lens fitting. Eye Contact Lens. 2011 Jan;37(1):20-5. doi: 10.1097/ICL.0b013e3182048fb9. PMID 21178696
- [Background] Morgan PB, Efron N, Woods CA; International Contact Lens Prescribing Survey Consortium. An international survey of toric contact lens prescribing. Eye Contact Lens. 2013 Mar;39(2):132-7. doi: 10.1097/ICL.0b013e318268612c. PMID 23392302
- [Background] Efron N, Nichols JJ, Woods CA, Morgan PB. Trends in US Contact Lens Prescribing 2002 to 2014. Optom Vis Sci. 2015 Jul;92(7):758-67. doi: 10.1097/OPX.0000000000000623. PMID 26101823
- [Background] Richdale K, Berntsen DA, Mack CJ, Merchea MM, Barr JT. Visual acuity with spherical and toric soft contact lenses in low- to moderate-astigmatic eyes. Optom Vis Sci. 2007 Oct;84(10):969-75. doi: 10.1097/OPX.0b013e318157c6dc. PMID 18049362
- [Background] Cox SM, Berntsen DA, Bickle KM, Mathew JH, Powell DR, Little BK, Lorenz KO, Nichols JJ. Efficacy of Toric Contact Lenses in Fitting and Patient-Reported Outcomes in Contact Lens Wearers. Eye Contact Lens. 2018 Sep;44 Suppl 1:S296-S299. doi: 10.1097/ICL.0000000000000418. PMID 28945646
- [Background] Woods J, Woods CA, Fonn D. Early symptomatic presbyopes--what correction modality works best? Eye Contact Lens. 2009 Sep;35(5):221-6. doi: 10.1097/ICL.0b013e3181b5003b. PMID 19675462
- [Background] Morgan PB, Efron SE, Efron N, Hill EA. Inefficacy of aspheric soft contact lenses for the correction of low levels of astigmatism. Optom Vis Sci. 2005 Sep;82(9):823-8. doi: 10.1097/01.opx.0000177792.62460.58. PMID 16189492
- [Background] Calabrese A, To L, He Y, Berkholtz E, Rafian P, Legge GE. Comparing performance on the MNREAD iPad application with the MNREAD acuity chart. J Vis. 2018 Jan 1;18(1):8. doi: 10.1167/18.1.8. PMID 29351351
- [Background] GRIZZLE JE. THE TWO-PERIOD CHANGE-OVER DESIGN AN ITS USE IN CLINICAL TRIALS. Biometrics. 1965 Jun;21:467-80. No abstract available. PMID 14338679
- [Background] Buckhurst PJ, Wolffsohn JS, Gupta N, Naroo SA, Davies LN, Shah S. Development of a questionnaire to assess the relative subjective benefits of presbyopia correction. J Cataract Refract Surg. 2012 Jan;38(1):74-9. doi: 10.1016/j.jcrs.2011.07.032. Epub 2011 Nov 10. PMID 22078121
- [Background] Thompson KA, Soler AP, Smith RM, Jarett L. Intranuclear localization of insulin in rat hepatoma cells: insulin/matrix association. Eur J Cell Biol. 1989 Dec;50(2):442-6. PMID 2697559
- [Background] Bhaskaran A, Babu M, Abhilash B, Sudhakar NA, Dixitha V. Comparison of smartphone application-based visual acuity with traditional visual acuity chart for use in tele-ophthalmology. Taiwan J Ophthalmol. 2022 May 13;12(2):155-163. doi: 10.4103/tjo.tjo_7_22. eCollection 2022 Apr-Jun. PMID 35813797
- [Background] Hazari H, Curtis R, Eden K, Hopman WM, Irrcher I, Bona MD. Validation of the visual acuity iPad app Eye Chart Pro compared to the standard Early Treatment Diabetic Retinopathy Study chart in a low-vision population. J Telemed Telecare. 2022 Oct;28(9):680-686. doi: 10.1177/1357633X20960640. Epub 2020 Sep 26. PMID 32985378
- [Background] Zhang ZT, Zhang SC, Huang XG, Liang LY. A pilot trial of the iPad tablet computer as a portable device for visual acuity testing. J Telemed Telecare. 2013 Jan;19(1):55-9. doi: 10.1177/1357633X12474964. Epub 2013 Feb 22. PMID 23434538
- See also: Howard, J. (2016, July 29). Americans Devote More than 10 Hours a Day to Screen Time, and Growing. — https://edition.cnn.com/2016/06/30/health/americans-screen-time-nielsen/index.html

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT06230263/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT06230263/ICF_001.pdf